CLINICAL TRIAL: NCT02710279
Title: Response to Social Rejection in Suicidal Behavior
Acronym: SADS-CS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties in recruitment
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9615; 2015-A01308-41 (Other: Agence Nationale de Sécurité des Médicaments)
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2021-12

CONDITIONS: Unipolar Depression
Keywords: Psychiatry; Depressive disorder; Suicide
MeSH Terms: conditions — Depressive Disorder; Suicide | interventions — Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Depressive patients (Other): Depressive patients with or without story of suicidal behavior will pass the TSST and will have a psychological assessment to complete with a questionnaire on their smartphone
  Interventions: Behavioral: Trier Social Stress Test (TSST); Device: smartphone

INTERVENTIONS:
Behavioral: Trier Social Stress Test (TSST) — For the TSST the participants are instructed to imagine having applied for their "dream job" and that they are now invited to a job interview. Three successive phases: (1) A preparation period (3 min), (2) a free speech: explain why you are the best candidate for the job (5 min), (3) a mental arithmetic complex task (5 min). The two tasks (task 2 and 3) are performed in front of a selection committee, three persons dressed in white lab coats, acting in a reserved manner and providing no facial or verbal feedback. Additionally, participants are told that they are video-taped and told that their performance will be evaluated. (in fact, there is no video-tape, just a false camera). After the TSST, patients have to answer to a questionnaire on their smartphone, 5 times a day during 7 days.
Device: smartphone

SUMMARY:
Suicide is a major health problem that causes annually a million death worldwild. In the stress-vulnerability model, suicidal behavior (SB) results from the interaction between an individual's predisposition and stressful condition. We hypothesized that the sensitivity to social exclusion may represent a core component of the suicidal vulnerability Recent evidence also suggest that inflammatory mediators plays a critical role in SB. Furthermore, social stressors are particulary strong and specific triggers of inflammatory response.

To sum up, patients carrying a suicidal vulnerability are expected to present greater responses to social rejection in terms of inflammatory activity and psychological pain.

The aim of the study is to evaluate the psychological and inflammatory responses to a social stressor validated, the Trier Social Stress Test (TSST) . We will also investigate the moderating effect of childhood abuse, attachment, trait rejection sensitivity and social isolation.

In the second part of the study, we will also investigate the prospective association between inflammatory responses induces by laboratory paradigms of social rejection and the occurrence of social distress, suicidal ideation and psychological pain in response to social exclusion events in real life (using ecological momentary assessment).

DETAILED DESCRIPTION:
Over one year, we will recruit 140 female outpatients suffering from a major depressive episode with (n=70) and without any history of suicide attempt (n=70) from a specialized clinic for mood disorders and SB.

First visit: clinical, biological and neuropsychological assessment Second visit: The TSST is a standardized laboratory psychosocial stress protocol that involves public speaking, role play, and mental arithmetic tasks in front of a panel of confederate judges. Blood samples will be obtained before the introduction to the TSST and immediately after and at + 30, + 60, + 90, and + 120 min. Self-ratings of emotional states, anxiety, anger and psychological pain will be completed at the same times.

Third visit: Participants will be instructed to carry a smartphone with them for one week, and to record at each alarm signal daily life events, negative emotions, psychological pain, suicidal ideas, and specific attributions to these events. Participants will be signalled five times a day during the period. Subjects will be contacted by telephone halfway through the assessment period to monitor and encourage compliance.

ELIGIBILITY:
Inclusion Criteria:

* Non specifics
* Female
* Between 18 and 65 years
* Main diagnosis of unipolar major depressive episode (DSM-IV criteria)
* Having signed informed consent
* Able to understand nature, aims, and methodology oh the study
* Specifics :
* Having a personal history of suicidal behavior (group : depressed patient with history of SB) OR
* Not Having personal history of suicidal behavior (group : depressed patient without history of SB)

Exclusion criteria:

* Inflammatory or intercurrent pathology
* Lifetime history of schizophrenia, or schizoaffective or bipolar disorder, according to DSM-IV criteria;
* Current diagnosis of substance abuse or dependence in the last year (excluding tobacco)
* Current organic mental disorder or mental retardation, or severe comorbid medical condition
* Participation in another clinical trial
* Pregnancy
* Not able to speak, read and understand French
* Patient on protective measures (guardianship or trusteeship)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Psychological pain response to Trier Social Stress Test (TSST) assessed by visual analogic sale | up to one week
  comparaison of psychological pain response between group with personal history of suicid attempt and group without personal history of suicid attempt

SECONDARY OUTCOMES:
Inflammatory response to TTST | up to one week
  comparaison of blood markers of inflammation between groups
Impact of loneliness and childhood abuse on inflammatory markers | up to one week
  comparaison of sacles scores (ESUL : loneliness scale and CTQ : childhood abuse scale) between groups on inflammatory markers
impact of neuropschychological function on psychological pain | up to one week
  comparaison of neuropsychological tests between groups on psychological pain assessed by visual analogic scale
Social rejection assessed by likert scale in real life condition with a smartphone | 7 days after the TSST
  comparaison between groups whether inflammatory / psychological pain reactivity to a single experimental episode of social rejection in the laboratory relates to real-world social experience. It consists on self-assessments (with a smartphone) by Likert scales (feelings of social disconnection or rejection during their most recent social interaction, mood, negative affects, suicidal ideation, psychological pain), 5 times per day during 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Courtet, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided